CLINICAL TRIAL: NCT02760108
Title: Parkinson's Families Project
Acronym: PFP
Status: Recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: Parkinson's UK (Other); Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 14/0800
Record Dates: First submitted 2016-04-22; First posted 2016-05-03 (Estimated); Last update posted 2019-06-12 (Actual); Status verified 2019-06

CONDITIONS: Parkinson's Disease; Parkinsonism
Keywords: Early onset Parkinson's disease; Familial Parkinson's disease; Parkinson's disease; Genetics
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — DNA will be extracted from whole blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Index case: Patients with a family history of Parkinson's/parkinsonism, and/or early onset Parkinson's/parkinsonism. The first individual member from a family who is recruited to the study.
- Affected relatives: Patients with Parkinson's/parkinsonism who are first or second degree relatives of an Index Case.
- Unaffected relatives: Participants who do not have Parkinson's/parkinsonism and are first or second degree relatives of an Index Case.

SUMMARY:
One person in every 500 has Parkinson's and around 127,000 people are living with the condition in the UK. The aim of the study is to identify new genes that predispose or cause Parkinson's Disease or Parkinsonism. There is a pressing need to study the genetic makeup of family members both with and without Parkinson's. As families share a common genetic background, it is easier to find new Parkinson's genes by studying the genetic makeup of people with Parkinson's alongside other members of their families. We are particularly interested in studying the genetic makeup of two groups of people:

1. those who developed Parkinson's before the age of 45; and
2. those who have a family history of other relatives affected by Parkinson's.

By identifying genetic factors that cause Parkinson's, we hope to understand more about the condition. Doing so will lead to the development of better diagnosis, improved disease models, and we hope in time, to the development of better treatment.

DETAILED DESCRIPTION:
One person in every 500 has Parkinson's and around 127,000 people are living with the condition in the UK. Unfortunately, it is a progressive disease that has no cure. Many treatments are available that can improve or maintain someone's quality of life, but the investigators would like to develop treatments that can be used much earlier in the disease process. These could slow down the disease or prevent it from progressing further.

For most people who develop Parkinson's there is no clear underlying cause. However, the investigators are particularly interested in the minority of people diagnosed with Parkinson's who have either early onset disease and/or other relatives affected with Parkinson's. The investigators believe that variations in inherited material (genes) can sometimes cause the disease, and this may run in families. This opens the door to a range of studies on the effects of gene variation at a nerve cell and brain level, which the investigators hope will lead to new targeted treatments.

It is already known that some rare gene variants can cause Parkinson's. Some of these are inherited in what is called an 'autosomal dominant' way i.e. each child of a person with this type of gene change has a 50% chance of inheriting it. However, it is also known that not everyone who carries the change will go on to develop the disease. Some people appear to be protected against developing the disease and the investigators would like to understand this better. Other variants, particularly important in early onset Parkinson's are "recessive", and in this form of inheritance there is a very low risk to parents and children.

The investigators are looking closely at the genetic makeup of people with Parkinson's in comparison with unaffected people and in comparison to unaffected and affected family members in order to find out more about which gene changes can cause Parkinson's.

Following the identification of genetic variation that causes Parkinson's, in collaboration with the NHS and other researchers, the investigators plan to: 1) develop new NHS tests of Parkinson's and 2) develop new disease model which can act as a testbed for new treatments

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of Parkinson's disease or parkinsonism, and either family history of Parkinson's/parkinsonism (first or second degree family member affected by Parkinson's or parkinsonism) AND/OR Early onset Parkinson's/parkinsonism (symptom onset before the age of 45 years) First or second degree family member of an Index Case, affected or unaffected by Parkinson's/parkinsonism.

Aged over 16 years

Exclusion Criteria:

Lack of capacity to consent to participate in the project.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from specialist secondary care clinics at collaborating centres in the United Kingdom. Participants can also be recruited from the community, through advertisements in patient newsletters and websites.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-04; Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who are clinically affected by Parkinson's disease or Parkinsonism, in relation to genetic factors. | Through study completion, approximately 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Huw Morris, PhD, FRCP, Principal Investigator — University College, London
Locations (2):
- United Kingdom (2):
  - Royal Free London NHS Foundation Trust, London
  - University College London Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Anonymous study information may made available to collaborators at other sites in the UK and overseas and may be made publicly available to bona fide researchers to enable the combined analysis of samples from different, large patient series around the world. This may include commercial companies. These are rare conditions and it is likely that sharing and collaboration between research groups and companies in different countries will be needed to make the best use of the study. Transfer of study data will be managed in a highly secure and anonymised format.